CLINICAL TRIAL: NCT01158365
Title: Single Center, Open, Cross-over, Phase III Study for Comparative Evaluation of Safety Use and Efficacy in the Odor Reduce and Vaginal Moisturize Increase for Intimates Use Products Dermacyd Femina Delicata, Dermacyd Femina Breeze, Dermacyd Teen Sweet Flower, Dermacyd Teen Fresh Mix and Dermacyd Femina Comparing to the Control Product Glycerine Vegetal Soap Granado Traditional.
Brief Title: Dermacyd in Odor Reducing.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LACAC_L_05401; U1111-1115-3484 (Other: UTN)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (2):
- Dermacyd (different fragrances) (Experimental): Day 1 until 30: Investigational Product (Dermacyd) Day 31 until 37: wash-out Day 38 until 67: Glycerine Vegetal Soap Granado Traditional
  Interventions: Drug: LACTIC ACID (Dermacid); Drug: Glycerine Vegetal Soap Granado Traditional
- Glycerine Vegetal Soap Granado Traditional (Active Comparator): Day 1 until 30: Glycerine Vegetal Soap Granado Traditional Day 31 until 37: wash-out Day 38 until 67: Investigational Product (Dermacyd)
  Interventions: Drug: LACTIC ACID (Dermacid); Drug: Glycerine Vegetal Soap Granado Traditional

INTERVENTIONS:
Drug: LACTIC ACID (Dermacid) — Route of administration: local
Drug: Glycerine Vegetal Soap Granado Traditional — Route of administration: local

SUMMARY:
Primary Objective:

- To prove the efficacy superiority in reducing the genital odor and increase hydration in mucosa genital comparing the use of Dermacyd (different fragrances) and Glycerine Vegetal Soap Granado Traditional

Secondary Objective:

- To evaluate the safety in normal conditions of use, verifying clinical signs and lab exams.

ELIGIBILITY:
Inclusion criteria:

* Perfect mucosa in the product analysis region
* Volunteers with active sexual life: normal Papanicolau test performed less than one year is mandatory
* Bacterioscopy describing the vaginal flora
* Negative Trichomonas vaginalis test
* Negative Whiff test
* Willingness in using preservative in the sexual intercourse during the study period
* Use the same category cosmetics products
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion

Exclusion criteria:

* Use of antiinflammatory / immunosuppression / antihistaminic drugs
* Atopic or allergy history to cosmetic products
* Active cutaneous disease (local and/or disseminated) in the evaluated area
* Disease which can cause immunosuppression, such as diabetes, HIV, etc.
* Endocrine pathology such as thyroid disease, ovarian or adrenal gland disturbs
* Intense solar exposure (to get a tan) during the 15 days before the evaluation
* Gynecologic treatment until four weeks before the evaluation
* Any vaginal infection detected during the inclusion
* Other conditions considered by the investigator as reasonable for exclude the patient in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction of genital odor and increase hydration in genital mucosa | From the treatment start to the end of the study (day 67)
  Patient's questionnaire will be completed at V1, V2 and V4. Reduction of vaginal odor, increase in the moisture area, and perception about some items like foam, facility of rinsing, final touch of the mucosa, final fragrance, and cleaning sensation will be rated on a 5-point scale.

SECONDARY OUTCOMES:
Evaluation of the integrity of the mucosa | From the treatment start to the end of the study (day 67)
  Onset of erythema, edema, scaling, blisters or other clinical sign will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Investigational Site Number 076-001, Osasco, Brazil